CLINICAL TRIAL: NCT07231315
Title: INTEnsive Ambulance-delivered Blood Pressure Reduction in Biomarker-identified Hyper-ACute Intracerebral Haemorrhage Trial - Validation Study
Brief Title: INTERACT4 Expansion - Validation Study
Acronym: INTERACT4 Exp
Status: Not yet recruiting | Type: Observational
Sponsor: The George Institute (Other)
Responsible Party: Sponsor
Other Study IDs: P01720
Record Dates: First submitted 2025-09-17; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: LVOne — LVOne is an in vitro diagnostic rapid lateral flow chromatographic immunoassay kit

SUMMARY:
As an investigator-initiated and conducted, multi-centre, open-label, single-arm prospective observational trial, INTERACT4 Expansion aims to evaluate the diagnostic accuracy of GFAP measured using a point-of-care device, for identifying ICH in participants presenting with acute stroke-like symptoms in the pre-hospital setting compared with imaging-confirmed ICH.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age ≥18 years);
2. Acute syndrome that is due to presumed acute stroke, defined as FAST (Face, Arm, Speech, Time) scores of ≥2 with an arm motor deficit;
3. Time ≤3 hours from last seen well;
4. Systolic BP (SBP) ≥150mmHg.

Exclusion Criteria:

1. Participants in coma (no response to tactile/verbal stimulation); or/and do not respond to "P" or "U" on the alert/verbal/painful/unresponsive (APVU) responsiveness scale;
2. Severe known co-morbid disease (e.g. cancer, chronic airflow disease, severe dementia, severe heart failure, pre-existing disability [needing help]);
3. Known history of epilepsy or seizure at onset;
4. Recent head injury (where there is potential for another type of intracranial haemorrhage or head trauma);
5. Hypoglycaemia (glucose<4.0 mmol/L) as measured in the ambulance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected acute stroke presenting to ambulance services
Sampling Method: Non-Probability Sample
Enrollment: 465 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants without ICH on hospital-based brain CT who are correctly identified as negative based on GFAP point-of-care measurement. (Specificity) | From enrolment to initial CT scan up until 7 day assessment

SECONDARY OUTCOMES:
Proportion of participants with ICH on hospital-based brain CT who are correctly identified as positive based on GFAP point-of-care measurement. | From enrolment to initial CT scan up until 7 day assessment
Proportion of participants with a positive GFAP point-of-care measurement who are confirmed to have ICH on hospital-based brain CT. | From enrolment to initial CT scan up until 7 day assessment
Proportion of participants with a negative GFAP point-of-care measurement who are confirmed to not have an ICH on hospital-based brain CT. | From enrolment to initial CT scan up until 7 day assessment
Feasibility of recruitment, assessed by the proportion of enrolled participants over the number of stroke calls in the participating networks during the study period. | From enrollment to end of the study.
Feasibility of protocol delivery, assessed by the proportion of participants for whom all required study assessments in the ambulance were completed among those in whom assessments were initiated. | From enrolment to transfer to hospital at day 1
  Study assesments include: participant screening, GFAP testing with the point-of-care device, and data entry
Feasibility of GFAP testing in the prehospital setting, defined as the proportion of enrolled participants in whom GFAP testing was successfully completed using the point-of-care device in the ambulance. | From enrolment to transfer to hospital at day 1
Correlation of GFAP measurement by the point-of-care device against a laboratory assay. | From enrolment to transfer to hospital at day 1

OTHER OUTCOMES:
Sensitivity, specificity, positive predictive value, and negative predictive value for identifying ICH using a (+) GFAP combined with a (-) D-dimer result on the point-of-care device, compared with hospital-based brain CT. | From enrolment to initial CT scan up until 7 day assessment
  Exploratory outcome

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Liverpool Hospital, Sydney, New South Wales
  - Nepean Hospital, Sydney, New South Wales
  - New South Wales Ambulance, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: Undecided